CLINICAL TRIAL: NCT05350956
Title: A Prospective, Multi-cohort, Open-label Clinical Study of the Efficacy and Safety of Herombopag in Tumors-associated Thrombocytopenia
Brief Title: A Clinical Study of Herombopag in Tumors-associated Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hong Zong, The First Affiliated Hospital of Zhengzhou University, Oncology Department， Chief Physician, The First Affiliated Hospital of Zhengzhou University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HQBP-ZH-001
Record Dates: First submitted 2022-03-29; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Tumor Therapy-related Thrombocytopenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herombopag monotherapy (Experimental)
  Interventions: Drug: TPO-RA (Herombopag)
- Herombopag is treated in combination with rhTPO(Recombinant human thrombopoietin) (Experimental)
  Interventions: Drug: TPO-RA (Herombopag) and rhTPO(Recombinant human thrombopoietin)

INTERVENTIONS:
Drug: TPO-RA (Herombopag) — During the correction period, subjects will receive a dose of Herombopag starting at 5-7.5mg once daily, orally for 14 days, subject to dosing adjustment (or discontinuation) depending on their platelet response or at the investigator's discretion. In the secondary prophylaxis phase, Herombopag 5mg once daily, starting 5 days before antineoplastic therapy and continuing for 10-14 days.
  Arms: Herombopag monotherapy
Drug: TPO-RA (Herombopag) and rhTPO(Recombinant human thrombopoietin) — During the correction period, subjects will receive a combination of Herombopag and rhTPO, Herombopag starting at a recommended dose of 5mg once daily for 14 days. The recombinant human thrombopoietin dose is 300U/kg. bw/day or 15000U/day per person, once daily, for 14 consecutive days (or as determined by the investigator). In the secondary prophylaxis phase, Herombopag 5mg once daily, starting 5 days before antineoplastic therapy and continuing for 10-14 days.
  Arms: Herombopag is treated in combination with rhTPO(Recombinant human thrombopoietin)

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Herombopag in tumors-associated thrombocytopenia

DETAILED DESCRIPTION:
CIT is one of the most common complications of tumor treatment, which is caused by the inhibition of anticancer chemotherapy drugs on megakaryocytes in bone marrow, resulting in platelet count lower than 100×109/L in peripheral blood, and is a common hematological toxic reaction in clinic. CIT leads to an increased risk of bleeding and transfusion, and severe CIT can cause intracranial bleeding and death. The use of platelet infusion is limited and ineffective in 25% of patients. rhIL-11 increases the incidence of cardiovascular events and rhTPO may produce immunogenicity. Currently, TPO-RA is recommended for the treatment of CIT by consensus guidelines at home and abroad. The study was designed to explore the safety and efficacy of Herombopag in the treatment of tumour-associated thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, no gender limitation;
2. Participants with solid tumors confirmed by histopathological or cytological examination;
3. During the current tumor treatment cycle, the participants whose PLT<50×109/L, and will receive the current tumor treatment regimen for at least 1 cycle;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
5. Voluntarily participated in the study and signed the informed consent with good compliance.

Exclusion Criteria:

1. Suffering from any of the following diseases of the hematopoietic system other than thrombocytopenia caused by tumor therapy, including but not limited to leukemia, primary immune thrombocytopenia, myeloid proliferative disease, multiple myeloma and myelodysplastic syndrome;
2. Suffering from thrombocytopenia (not caused by tumor treatment), including but not limited to chronic liver disease, hypersplenism, infection, and bleeding, within 6 months prior to screening;
3. Bone marrow invasion or bone marrow metastasis;
4. Received radiation therapy to the pelvis, spine and bone field within 3 months prior to screening; or is/is expected to receive radiation therapy.
5. Received TPO-RA drugs (such as altrepopal and romistine), or rhTPO or rhIL-11 in the current cancer treatment cycle;
6. Received platelet transfusion within 3 days prior to randomization;
7. Participants with known or expected allergy or intolerance to the active ingredient or excipient of Herombopag Olamine tablets;
8. Pregnant or lactating women;
9. Participants who are participating in other clinical trials.
10. Other conditions that the investigator determines are not suitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
During the correction period, the percentage of patients whose platelets returned to normal within 14 days | up to 14 days
  Percentage of patients whose platelets returned to normal within 14 days

SECONDARY OUTCOMES:
During the correction period, the median time for platelet values to return to normal | up to 60 days
  Median time for platelet values to return to normal
During the correction period, the Median time for platelet count to return to 75×109/L | up to 60 days
  Median time for platelet count to return to 75×109/L
During the correction period, the median time for platelet count to return to 50×109/L | up to 60 days
  Median time for platelet count to return to 50×109/L
During the correction period, the percentage of patients whose platelets returned to75×109/L within 14 days | up to 14 days
  Percentage of patients whose platelets returned to75×109/L within 14 days
During the correction period, the percentage of patients whose platelets returned to 50×109/L within 14 days | up to 14 days
  Percentage of patients whose platelets returned to 50×109/L within 14 days
During the correction period, platelet infusion rate after initiation of Herombopag therapy. | up to 14 days
  During the correction period, platelet infusion rate after initiation of Herombopag therapy.
During the prophylaxis period, the proportion of patients whose PLT<75×109/L | up to 14 days
  During the prophylaxis period, the proportion of patients whose PLT<75×109/L
During the prophylaxis period, the proportion of patients whose PLT<50×109/L | up to 14 days
  During the prophylaxis period, the proportion of patients whose PLT<50×109/L
During the prophylaxis period, platelet counts are at their lowest. | up to 14 days
  During the prophylaxis period, platelet counts are at their lowest.
During the prophylaxis period, platelet infusion rate after initiation of Herombopag therapy. | up to 14 days
  During the prophylaxis period, platelet infusion rate after initiation of Herombopag therapy.
Platelet value curve | up to 60 days
  Platelet value curve

CONTACTS AND LOCATIONS:
Overall Officials: Zong Hong, Professor, Principal Investigator — The First Affiliated Hospital of Zhengzhou University